CLINICAL TRIAL: NCT02272309
Title: Neurophysiological Assessment of Healthy and Impaired Human Lower Urinary Tract Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrich Mehnert (Other)
Responsible Party: Sponsor-Investigator, Ulrich Mehnert, Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH_2013-0518/PB_2016-00498
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Healthy volunteers (Experimental): Healthy volunteers
  Interventions: Procedure: EEG and EP measurement
- Patients with LUTS (Experimental): Patients with LUTS
  Interventions: Procedure: EEG and EP measurement
- Patients with LUTS and treatment (Experimental): Patients with LUTS and treatment
  Interventions: Procedure: EEG and EP measurement

INTERVENTIONS:
Procedure: EEG and EP measurement

SUMMARY:
Study part 1 will consist of sensory evoked cortical potential (SEP) measurements of the lower urinary tract (LUT) in healthy subjects using different stimulation frequencies from 0.25 to 3Hz to find the most effective frequency in regard to acquisition time for reliable SEP response rates. Study part 2 will consist of a series of consecutive SEP measurements in patients with LUT symptoms during low bladder volume and maximum cystometric capacity to assess reliability of measurements and influence of potential concomitant LUTS treatments.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers:

* Written informed consent,
* good mental and physical health,
* age >18y,

Patients with LUTS and Patients with LUTS and treatment:

* Written informed consent,
* age >18y,
* prior urodynamic investigation,
* LUTS since >6months with or without detrusor overactivity

Exclusion Criteria:

healthy volunteers:

* any neurological or urological pathology,
* current pregnancy or lactation,
* urinary tract infection,
* hematuria,
* any previous pelvic or spine or craniocerebral surgery,
* any anatomical anomaly of the LUT or genitalia,
* any metabolic disease,
* any LUT malignancy,
* bladder capacity <150mL,
* SDV at 60mL;

Patients with LUTS and Patients with LUTS and treatment:

* current pregnancy or lactation,
* urinary tract infection,
* gross hematuria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
N1latency of LUT SEPs | 2-3 measurements within 4-16 weeks from first exam

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liechti MD, van der Lely S, Knupfer SC, Abt D, Kiss B, Leitner L, Mordasini L, Tornic J, Wollner J, Mehnert U, Bachmann LM, Burkhard FC, Engeler DS, Pannek J, Kessler TM. Sacral Neuromodulation for Neurogenic Lower Urinary Tract Dysfunction. NEJM Evid. 2022 Nov;1(11):EVIDoa2200071. doi: 10.1056/EVIDoa2200071. Epub 2022 Jul 7. PMID 38319849
- [Derived] van der Lely S, Stefanovic M, Schmidhalter MR, Pittavino M, Furrer R, Liechti MD, Schubert M, Kessler TM, Mehnert U. Protocol for a prospective, randomized study on neurophysiological assessment of lower urinary tract function in a healthy cohort. BMC Urol. 2016 Nov 25;16(1):69. doi: 10.1186/s12894-016-0188-9. PMID 27887601